CLINICAL TRIAL: NCT04502511
Title: Heterogeneity of Critical Illness: Exploring New Risk Factors for Severity of Disease in Intensive Care Patients. A Cohort Study
Brief Title: Heterogeneity of Critical Illness: a Cohort Study
Acronym: HEALICS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Frederik Keus, Principal investigator, University Medical Center Groningen
Other Study IDs: 202000405
Record Dates: First submitted 2020-07-27; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Critically Ill; Organ Failure, Multiple
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult critically ill patients in the ICU: Acutely admitted to the ICU
  Interventions: Diagnostic Test: Standard diagnosis test

INTERVENTIONS:
Diagnostic Test: Standard diagnosis test — Care as usual

SUMMARY:
Rationale: There is large heterogeneity in disease states of critically ill patients at ICU admittance and there is also large heterogeneity in their disease severity during ICU stay. Still, some patients may show remarkable similarities in disease patterns. There is a lack of understanding of causal mechanisms that lead to divergent outcomes in critically ill patients, and at the same time different diseases may share common underlying, yet unidentified, causal pathways that could explain similarities between different diseases.

Objective: To explore the association between patient characteristics and the severity of organ failure in critically ill patients admitted to the ICU Study design: Prospective cohort study Study population: Adult critically ill patients in the ICU Intervention (if applicable): not applicable Main study parameters/endpoints: Maximum severity of organ failure observed during ICU stay measured by the maximum SOFA score and quality of life at one year follow-up

DETAILED DESCRIPTION:
Nature and extent of the burden and risks associated with participation, benefit and group relatedness: <All patients will undergo physical examination, including ultrasound evaluation upon ICU admission according to standard practice care. The burden will be a blood sample (and urine sample) at admission. Blood sample will be obtained by arterial line (or venous access) which is part of standard ICU care. So there will be no additional puncture for this study. Collection of variables during ICU stay will all be either part of standard clinical care or include extra physical examination or ultrasound evaluation. For follow-up patients will be evaluated by phone at 6 months and at 12 months by home-visit. This is also already part of the investigator's evaluation of quality of care. Except for blood sampling, all study related procedures have previously been approved by the Institutional Review Board (IRB). The patient will experience no individual benefit.

ELIGIBILITY:
Inclusion Criteria:

* Adults Definition: age ≥18 years.
* Emergency admission to the ICU Definition: patients who are acutely admitted to the ICU due to acute or unexpected critical illness, either from the emergency department or the ward or transferred from an ICU (or a ward) from another hospital.

Exclusion Criteria:

* Planned admission
* Absence of an invasive arterial or venous line for blood sampling.
* Any continued cardiopulmonary resuscitation efforts upon admission which limit access to the patient for research activities.
* Main ICU admission reason chronic (non-invasive) home ventilation
* Main ICU admission reason normothermic treatment after cardiac arrest
* Main ICU admission reason ischemic stroke, intracerebral bleeding, or isolated neurotrauma
* Main ICU admission reason Coronavirus Disease 2019 (COVID-19)
* Solid organ or hematopoietic stem cell transplant during current hospital admission
* Strict isolation due to any contagious disease
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients acutely admitted to the ICU
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Severity of organ failure observed during ICU stay | During ICU admission with a maximum of 90 days
  The primary prognostic outcome will be the maximum SOFA score during ICU stay. The daily maximum SOFA score will be considered up to a maximum of 90 days.

SECONDARY OUTCOMES:
Follow-up Quality of life data | 6 and 12 months after ICU discharge
  Patients will be evaluated by questionnaires at 6 and 12 months follow-up.Follow-up data will include survival status and data on quality of life.
  * Patients psychological functioning will be evaluated using the Short Form 20 and the Hospital Anxiety and Depression Scale (HADS).
  * Patients physical functioning data will be measured by the KATZ ADL index and the Clinical Frailty Score. In addition, the Euro-Qol (EQ-5d) will be used.
  * Social functioning data will be collected using the General Functioning 6 scale (GF6) which is a subscale of the GF12 and is a quick and effective tool to assess the overall functioning of families. Data will be collected from both patients and family members. Return to work will only be evaluated at 12 months follow-up by 4 extra questions concerning the patients return to work.
  In addition we will explore and validate extended modifications on the total and domain level of the organ failure assessment score (SOFA+).

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Keus, PhD, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol
Time Frame: In two years
Access Criteria: On request

REFERENCES:
- [Derived] van der Aart TJ, Luxen M, Koeze J, Londen MV, Hackl M, Ter Maaten JC, van Meurs M, Bouma HR; the Acutelines research group. Validation of plasma microRNAs as biomarkers in sepsis associated acute kidney injury upon first clinical presentation reveals limited diagnostic and prognostic performance. PLoS One. 2025 Sep 4;20(9):e0331442. doi: 10.1371/journal.pone.0331442. eCollection 2025. PMID 40906653